CLINICAL TRIAL: NCT04429893
Title: Effectiveness of Adding Magnesium Sulphate to Bupivicaine in Ultrasound Guided Serratus Anterior Plane Block in Patients Undergoing Modified Radical Mastectomy
Brief Title: Magnesium Sulphate to Bupivicaine in Serratus Anterior Plane Block in Modified Radical Mastectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0304543
Record Dates: First submitted 2020-06-08; First posted 2020-06-12 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Cancer Breast; Chronic Pain Syndrome
Keywords: serratus anterior plane block; magnesium sulphate
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group BM (Experimental): The patients will receive 20 ml of 0.5% bupivacaine plus 150 mg magnesium sulphate in 0.9% normal saline with a total volume of 25 ml.
  Interventions: Drug: magnesium sulphate; Drug: bupivicaine
- Group B (Active Comparator): The patients will receive 20 ml of 0.5% bupivacaine plus 5 ml 0.9% normal saline with total volume 25 ml
  Interventions: Drug: bupivicaine

INTERVENTIONS:
Drug: magnesium sulphate — assess the pain intensity of magnesium sulphate as an adjuvant to bupivacaine in serratus anterior plane block for modified radical mastectomy
  Arms: Group BM
Drug: bupivicaine — assess the pain intensity of magnesium sulphate as an adjuvant to bupivacaine in serratus anterior plane block for modified radical mastectomy

SUMMARY:
Modified radical mastectomy may be associated with severe post-operative pain, leading to chronic pain syndrome which usually requires optimal perioperative pain management.

DETAILED DESCRIPTION:
Patients will be randomly into two equal groups (40 patients each) according to the adjuvant added to the local anesthetic (bupivacaine) in the serratus anterior plane block using a computer-generated random numbers concealed in sealed opaque envelopes. Group B: The patients will receive 20 ml of 0.5% bupivacaine plus 5 ml 0.9% normal saline with total volume 25 ml. Group BM: The patients will receive 20 ml of 0.5% bupivacaine plus 150 mg magnesium sulphate in 0.9% normal saline with a total volume of 25 ml.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients
* American Society Of Anesthesiologists (ASA) class I or II
* scheduled for elective unilateral modified radical mastectomy

Exclusion Criteria

* patient refusal
* bilateral breast surgery
* coagulation disorders
* body mass index> 35
* allergy to local anaesthetics or magnesium sulphate
* severe respiratory or cardiac disorders
* pre-existing neurological deficits
* liver or renal insufficiency

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
assessment of the pain intensity | 24 hours
  Pain assessment by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab Abd Elraof Abd Elaziz, Alexandria, Smouha, Egypt